CLINICAL TRIAL: NCT05318079
Title: Telehealth Virtual Reality Exergaming and Peer Networking Among People With Spinal Cord Injury
Brief Title: Telehealth Virtual Reality Exergaming for Spinal Cord Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not selected for funding.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Byron Lai, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300008605
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group virtual reality gaming (Experimental): The intervention will include home-based exercise using the Oculus Quest 2. Participants will be prescribed two gaming goals to achieve across the 8-week intervention. The first goal will be to play with the Quest for at least ≥60 minutes, 5 days per week (Monday - Friday) across the 8-week intervention: a total of 300 minutes. Participants can achieve these goals through either single- or multiplayer gaming but will be prescribed to engage in online multiplayer or peer-to-peer gaming at least 2 days per week.
  Interventions: Behavioral: Virtual Reality Gaming
- Wait-list Control (No Intervention): People who are randomized to the waitlist group will undergo 4-weeks of wait (habitual daily activities), followed by 8-weeks of VR intervention. People in the wait-group will be in the study for a total of 12 weeks.

INTERVENTIONS:
Behavioral: Virtual Reality Gaming — Peer-to-peer gaming.
  Arms: Group virtual reality gaming

SUMMARY:
This pilot feasibility study aims to test whether youth and adults with spinal cord injury can use a group virtual reality gaming intervention to exercise. A second purpose is to examine whether there are potential benefits to cardiometabolic health and psychosocial health.

DETAILED DESCRIPTION:
There are three purposes to this study.

The first purpose is to quantify feasibility through telemonitored exercise data: total play time, moderate exercise time, playtime with others, and compliance to the data collections. These variables will be compared against a priori criteria for acceptability. These variables will help determine whether modifications to the intervention protocol are necessary.

The second purpose is to qualitatively interview participants to explain underlying behavioral mechanisms that affect their participation in the program. This information will be used to explain how to improve implementation issues identified in Aim 1.

The third aim is to explore the potential effects of the program on self-reported psychosocial health and quality of life, hand-grip strength, and cardiometabolic health (blood cholesterol, lipids, pressure, and insulin) measured via home dried blood spot test.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of traumatic spinal cord injury (determined by International Classification of Disease [ICD] codes)
* a caregiver to support the participant if the participant is a child (<18 years of age)
* access to a Wi-Fi Internet connection in the home

Exclusion Criteria:

* physically active (defined as >150 minutes per week of moderate-to-vigorous intensity exercise in a typical week)
* cannot use the arms for exercise or operate the controller buttons using their fingers
* complete blindness or deafness
* recent myocardial infarction or electrocardiography changes, complete heart block, acute congestive heart failure, unstable angina, and uncontrolled severe hypertension [BP >/= 180/110 mmHg]
* prone to seizures

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Total play time | Intervention Week 1 - Week 8
  Percentage of the 300 minutes of prescribed play per week across the intervention.
Total exercise time | Intervention Week 1 - Week 8
  Moderate exercise minutes where prescription was met (percent of prescription achieved: weeks where the ≥90 minutes of moderate intensity exercise per week was achieved across the intervention, divided by total weeks).
Playtime with others | Intervention Week 1 - Week 8
  Measured by the number of play sessions with other players (online multiplayer and/or peer-gaming). This number will be totaled across the 8-week intervention and divided by 16 (the exercise prescription of 2 x per week of multiplayer gaming).
Compliance to baseline data collection | Week 0
  Number of pre data collections completed, converted into a percentage dividing by the total possible.
Compliance to post data collections | Week 9
  Number of pre data collections completed, converted into a percentage dividing by the total possible.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Week 0, Week 5, Week 9
  The Hospital Anxiety and Depression Scale is a 14-item self-report measure that provides separate scores for anxiety and depression. Hospital Anxiety and Depression Scale is a common clinical measure that has strong psychometric properties. Scores range from 0 to 42, where a higher score represents a worse level of depression.
World Health Organization Quality of Life | Week 0, Week 5, Week 9
  The World Health Organization Quality of Life is a self-report questionnaire with 26 items that cover 5 dimensions: physical health (7 items); psychological health (6 items); social relationships (3 items); environment (8 items); and overall quality of life (2 items). Raw scores are calculated for each domain on a lilkert scale of 1-5 (low domain score of 3, max domain raw score of 40. Raw scores are then multiplied by 4 to transform the raw score into a scaled score. Higher scores represent higher perceived ratings of quality of life.
Functional Grip Strength | Week 0, Week 5, Week 9
  Grip strength will be measured as an indicator of global muscular strength, using a low-cost hand-held dynamometer.
Critical factors that affected adherence | Intervention Week 9
  Participants will undergo one-on-one, semi-structured interviews after the intervention to identify critical factors that affected their participation to the intervention.
Changes in blood pressure | Week 0, Week 5, Week 9
  Changes in resting home-blood pressure (systolic and diastolic ) measured via blood pressure cuff across the intervention.
Changes in high sensitivity C-reactive protein (hsCRP) | Week 0, Week 5, Week 9
  Changes in high sensitivity C-reactive protein measured via blood spot test across the intervention.
Changes in hemoglobin A1c | Week 0, Week 5, Week 9
  Changes in hemoglobin A1c measured via blood spot test across the intervention.
Changes in fasting insulin | Week 0, Week 5, Week 9
  Changes in fasting insulin levels measured via blood spot test across the intervention.
Changes in fasting triglycerides | Week 0, Week 5, Week 9
  Changes in fasting triglycerides levels measured via blood spot test across the intervention.
Changes in total cholesterol | Week 0, Week 5, Week 9
  Changes in total cholesterol measured via blood spot test across the intervention.
Changes in low-density lipoprotein (LDL) | Week 0, Week 5, Week 9
  Changes in low-density lipoprotein via blood spot test across the intervention.
Changes in high-density lipoprotein (LDL) | Week 0, Week 5, Week 9
  Changes in high-density lipoprotein via blood spot test across the intervention.

IPD SHARING:
Plan to Share IPD: No